CLINICAL TRIAL: NCT03860987
Title: A Phase II Study of Neoadjuvant Androgen Deprivation Therapy Combined With Enzalutamide and Abiraterone Using Multiparametric MRI and 18F-DCFPyL-PET/CT in Newly Diagnosed Prostate Cancer
Brief Title: Neoadjuvant Androgen Deprivation Therapy Combined With Enzalutamide and Abiraterone Using Multiparametric MRI and 18FDCFPyL PET/CT in Newly Diagnosed Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 190062; 19-C-0062
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09-03

CONDITIONS: Castrate Sensitive Prostate Cancer
Keywords: Imaging; Prostatectomy; Anti-androgen Therapy; 18F-DCFPyL-PSMA
MeSH Terms: interventions — Goserelin; enzalutamide; abiraterone; 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Treatment
  Interventions: Drug: goserelin; Drug: Enzalutamide; Drug: Abiraterone; Drug: 18F-DCFPyL; Drug: Prednisone; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: goserelin — Goserelin will be administered SC at 10.8 mg every 12 weeks
Drug: Enzalutamide — Enzalutamide will be given orally at 160mg once daily
Drug: Abiraterone — Abiraterone will be taken orally at 1000 mg once daily
Drug: 18F-DCFPyL — 18F-labeled agent that is a high affinity small molecule inhibitor of PSMA to detect prostate cancer via PET imaging
Drug: Prednisone — Prednisone will be taken orally at 5mg twice a day for each dose, or 10 mg once a day. Doses should be taken about 12 or 24 hours apart
Procedure: Radical Prostatectomy — Radical Prostatectomy

SUMMARY:
Background:

Prostate cancer is a common cancer among men. There are several ways to treat it, including hormone blocking drugs, radiation therapy, and surgery. Researchers want to combine abiraterone and enzalutamide to see if there is a better way to treat prostate cancer. They also want to study a new radiotracer called 18F-DCFPyL, with the help of a scan called positron emission tomography/computed tomography (PET/CT) to see if there is a better way to detect prostate cancer.

Objective:

To develop improved techniques to localize and detect prostate cancer; and to develop new ways to treat prostate cancer

Eligibility:

Men ages 18 and older with prostate cancer that has not spread to other parts of the body

Design:

* Participants will have a medical evaluation to determine eligibility for the study.
* Participants will take three different medications daily by mouth and receive two injections during the course of the study.
* Participants will have a medical evaluation monthly (for 6 months) while taking the medications.
* Participants will have prostate MRI and PET/CT scans before treatment, 2 months after starting treatment and again before surgery. The radiotracer will be given by injection about 2 hours before the whole-body scan. The PET/CT scan itself is about an hour.
* Participants may be asked to do a biopsy before treatment and 2 months after starting treatment.
* Participants will have a full medical evaluation before surgery to remove their prostate.
* Participants will have a follow-up visit 3 months after surgery and then as needed.
* Participants will be contacted once a year for their PSA and testosterone levels for 5 years...

DETAILED DESCRIPTION:
Background:

* Most men diagnosed with prostate cancer will present with intermediate or high-risk disease, and many develop castrate resistant prostate cancer (CRPC) as curative strategies are often unsuccessful
* Treatment options typically involve radical prostatectomy (RP) or radiation therapy (RT) in combination with androgen deprivation therapy (ADT)
* PET imaging based on prostate specific membrane antigen (PSMA), including use of the radiotracer DCFPyL, which binds PSMA, has emerged as a sensitive modality to detect localized and metastatic prostate cancer
* It is unknown how androgen-targeted therapy affects expression of the androgen- regulated PSMA gene, FOLH1, and 18F -DCFPyL-PET/CT sensitivity; and, the correlation between response on 18F -DCFPyL-PET/CT imaging and clinical response needs further evaluation
* The use of highly effective androgen pathway inhibitors enzalutamide and abiraterone offers an opportunity to understand the characteristics of 18F -DCFPyL-PET imaging during treatment while potentially improving the cure rate of men with potentially lethal localized prostate cancer
* There remains a great need for improved techniques to determine mechanisms of treatment response and resistance

Objectives:

- To test the feasibility of 18F -DCFPyL-PET/CT for the localization of prostate cancer before, during, and after pre-operative treatment with ADT, enzalutamide, and abiraterone/prednisone in patients negative for metastatic disease

Eligibility:

* Pathologic diagnosis of castration-sensitive prostate cancer with intermediate- or high- risk features and no evidence of metastases beyond N1 on conventional imaging
* Candidates for radical prostatectomy
* Testosterone levels greater than or equal to 100 ng/dL
* ECOG PS 0-1
* Men age greater than or equal to 18 years

Design:

* Patients will be treated with ADT, enzalutamide, and abiraterone/prednisone for 6 months, followed by standard of care radical prostatectomy (RP)
* 18F-DCFPyL-PET/CT and mpMRI scans prior to treatment, during months 3-5 and after 6 months of treatment
* Prostate tumor biopsy (MR/US-guided) samples for research analyses at baseline and after mid-treatment imaging (post-month 2)
* It is anticipated that approximately 1.5 to 2 years may be required for accrual of up to 25 evaluable subjects.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histologically or cytologically confirmed prostate cancer confirmed by the Laboratory of Pathology, NCI, OR documented histopathological confirmation of prostate cancer from a CLIA-certified laboratory.
2. Must have previously untreated (with definitive therapy ie: surgery, systemic treatment or radiation therapy) prostate cancer with intermediate or high risk features defined as:

   * Intermediate risk (patient must have at least one of the features listed below):

     * PSA level is between 10 and 20 ng/ml,
     * Gleason score is 7, OR
     * Stage T2b or T2c,
   * High risk (patient must have at least one of the features listed below):

     * PSA > 20 at the time of diagnosis,
     * Gleason 8 or higher,
     * Seminal vesicle involvement,
     * Possible (on MRI) extra-capsular extension (T3 disease), OR
   * Clinical stage T4
3. Patients must be eligible for and must be planning to undergo radical prostatectomy
4. Patients must have testosterone levels greater than or equal to 100 ng/dL
5. Men age greater than or equal to18 years.

   Children are excluded because prostate cancer is not common in pediatric populations.

   Women are not eligible because this disease occurs only in men.
6. ECOG performance status 0-1.
7. Patients must have adequate organ and marrow function, and other laboratory parameters as defined below:

   * hemoglobin greater than or equal to 9 g/dL
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) less than or equal to 3 X institutional upper limit of normal
   * creatinine within normal institutional limits; OR,
   * creatinine clearance greater than or equal to 30 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (calculated via EGFR)
8. Lesions within prostate must be detectable on MRI for biopsy.
9. The effects of enzalutamide and abiraterone on the developing human fetus are unknown. For this reason and because androgen receptor antagonists as well as other therapeutic agents used in this trial are known to be teratogenic, male participants and their female partners of child bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence). Male participants should use a condom if having intercourse with a pregnant woman. Additionally, a condom plus another effective method of birth control is recommended during therapy and for 3 months after treatment for male participants having intercourse with a woman of reproductive potential. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately and her partner should inform the study team.
10. Ability of subject to understand and the willingness to sign a written informed consent document.
11. Willingness to adhere to protocol requirements (e.g., required biopsies).
12. Willingness to travel to NIH for follow-up visits.

EXCLUSION CRITERIA:

1. Patients who are receiving any other investigational agents (in the past 28 days) or herbal medications (within 1 day prior to registration).
2. Patients with evidence of distant metastatic disease beyond N1 (regional) lymph nodes on conventional imaging studies (e.g., CT, MRI or Bone Scan).
3. Patients who have received any prior definitive therapy (ie: surgery, systemic treatment or radiation therapy) for prostate cancer.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide, abiraterone or other agents used in study.
5. Clinically significant cardiac disease, e.g., New York Heart Association (NYHA) classes III-IV; uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension (greater than or equal to 160/100 mmHg on two consecutive readings), myocardial infarction in the previous 6 months as confirmed by an electrocardiogram (ECG).
6. Contraindication to biopsy:

   * Bleeding disorders for which a prostate biopsy would pose a bleeding risk
   * PT/PTT greater than or equal to 1.5 times the upper limit of normal
   * Artificial heart valve
7. Contraindication to MRI:

   * Patients weighing more than the weight limit or unable to fit the scanner
   * Allergy to MR contrast agent
   * Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic device
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
9. HIV-positive patients on antiretroviral therapy are ineligible because of potential pharmacokinetic interactions with study drugs. However, patients with long-standing (>5 years) HIV on antiretroviral therapy > 1 month (undetectable HIV viral load and CD4 count > 150 cells/microliter) may be eligible if the PI determines no anticipated clinically significant drug-drug interactions.
10. Patients undergoing active treatment for Hepatitis B or C infections.
11. Patients who have taken medications that are strong inhibitors or inducers of CYP3A4 or PgP within 14 days prior to enrollment and need to remain on these medications.
12. Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter PSA (e.g., phytoestrogens and saw palmetto) cannot be taken while patients are receiving enzalutamide and abiraterone.
13. Contraindication to steroid use.
14. Patients with malignancy within the past 3 years for which study drugs or a prostatectomy is a contraindication.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
disease status | 2 months
  The primary endpoint will be the disease status after completion of treatment relative to PSMA-PET imaging findings at 2 months

SECONDARY OUTCOMES:
pathological complete response rate | 5 years
  Evaluate the pathological complete response rate after neoadjuvant treatment with ADT, enzalutamide, and abiraterone/prednisone

CONTACTS AND LOCATIONS:
Overall Officials: Fatima H Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0062.html